CLINICAL TRIAL: NCT05154851
Title: An Expanded Access IND to Evaluate the Safety and Efficacy of Autologous HBadMSCs for the Treatment of a Single Pediatric Patient With Congenital Muscular Dystrophy.
Brief Title: HBCMD01- Expanded Access for the Treatment of Congenital Muscular Dystrophy.
Status: No longer available | Type: Expanded Access
Sponsor: Hope Biosciences Research Foundation (Industry)
Responsible Party: Sponsor
Other Study IDs: HBCMD01
Record Dates: First submitted 2021-12-09; First posted 2021-12-13 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-09

CONDITIONS: Congenital Muscular Dystrophy Due to Lamin A/C Mutation
Keywords: CMD; Muscular Dystrophy; Congenital; Stem cells; L-CMD
MeSH Terms: conditions — Muscular Dystrophy, Congenital, Lmna-Related; Muscular Dystrophies

STUDY DESIGN:
Expanded Access Types: Individual

INTERVENTIONS:
Biological: HB-adMSCs — HB-adMSCs (Hope Biosciences autologous adipose-derived mesenchymal stem cells) is manufactured by Hope Biosciences, L.L.C., a biotechnology company headquartered in Sugar Land, Texas.

SUMMARY:
This individual patient expanded access IND is requested for a patient diagnosed with LMNA-related congenital muscular dystrophy (L-CMD). In this expanded access, the patient will receive the investigational product through 14 intravenous infusions, followed by Follow-Up visit and an End of Study.

DETAILED DESCRIPTION:
This Expanded Access includes an up to 28 days screening period, a 44-week Treatment Period, and a 52-week Safety Follow-up Period. All periods are associated with evaluations and procedures that must be performed at specific time points.

-Screening

At the Screening Visit (Visit 1), the study's participant information will be collected by delegated personnel to evaluate trial eligibility. The following information is required to determine eligibility:

* Parent Permission before any trial-related activities.
* Collection of demographic information, such as age, race, ethnicity, date of birth, gender, and relevant medical and surgical history.
* Collection of Medical History and concomitant medications, including relevant information about study participants' past and present health.
* Inclusion and Exclusion criteria evaluation.
* Measurement of vital signs includes respiratory rate, body temperature, blood pressure, pulse rate, oxygen saturation, and weight and height measurement.
* Blood chemistry, Coagulation panel, Inflammatory Markers, & Hematology.
* Physical examination by Principal Investigator.

Within 28 days of the Visit 1 - Screening, the principal investigator must decide the participant's eligibility. Once the principal investigator has confirmed the subject's eligibility, the subject will be scheduled to receive Infusion 1.

Infusion 1 - Baseline

The following evaluations will be performed during this visit:

* Update medical history and concomitant medications if any change occurred since the last visit.
* Measure vital signs, including respiratory rate, body temperature, blood pressure, pulse rate, oxygen saturation, and weight measurement.
* Physical examination by Principal Investigator. As this 2-year-old is unable to walk or hold his head up without physical support, assessment for neurologic sequelae will include the following observations and discharge instructions for observations to continue at home by the primary caregivers:

  * Unusual /new weakness or numbness on one side of the body
  * New or different slurred speech or new language difficulty
  * New vision problems
  * Sudden lethargy or drowsiness
  * Seizure
* CHOP INTEND, PDMS-2 & PEDI-CAT by delegated personnel.
* Investigational product administration by delegated study personnel. HB-adMSCs should only be administered intravenously, with vital sign monitoring of two hours.
* Assess the incidence of any adverse event.
* Twenty-four hours after administration of the investigational product, study participants' parents or guardians will be contacted by telephone call to assess the incidence of adverse events.

  * Infusion 2 through Infusion 13.

The following assessments are necessary during these visits:

* Update medical history and concomitant medications if any change occurred since the last visit.
* Measure vital signs, including respiratory rate, body temperature, blood pressure, pulse rate, oxygen saturation, and weight measurement.
* Physical examination by Principal Investigator. As this 2-year-old is unable to walk or hold his head up without physical support, assessment for neurologic sequelae will include the following observations and discharge instructions for observations to continue at home by the primary caregivers:

  * Unusual /new weakness or numbness on one side of the body
  * New or different slurred speech or new language difficulty
  * New vision problems
  * Sudden lethargy or drowsiness
  * Seizure
* CHOP INTEND, PDMS-2 & PEDI-CAT by delegated personnel (at Inf. 1, 7, and EOS).
* Coagulation panel & Hematology. - (at Infusions 2,4,7,10, and EOS).
* Inflammatory Markers & Blood chemistry at Infusions 2, 7 and EOS.
* Investigational product administration by delegated study personnel. HB-adMSCs should only be administered intravenously, with vital sign monitoring of two hours.
* Assess the incidence of any adverse event.
* Twenty-four hours after administration of the investigational product, study participants' parents or guardians will be contacted by telephone call to assess the incidence of adverse events. The child's skin and eyes will be checked for symptoms of yellowing at each visit, and caregivers will be asked whether they have seen any vomiting, nausea, or the subject looking to be more tired than usual. Discharge instructions will include monitoring for these symptoms. Liver enzymes will be assessed at Screening, Infusion 2, 4, 7, 10, and End of Study per-protocol; however, these laboratory samples can be collected more often if the principal investigator indicates.

  * Safety Follow Up

The following evaluations will need to be completed during this visit:

* Update medical history and concomitant medications if any change occurred since the last visit.
* Measure vital signs, including respiratory rate, body temperature, blood pressure, pulse rate, oxygen saturation, and weight measurement.
* Physical examination by Principal Investigator.

  -End of Study Visit
* Update medical history and concomitant medications if any change occurred since the last visit.
* Measure vital signs, including respiratory rate, body temperature, blood pressure, pulse rate, oxygen saturation, and weight measurement.
* Collect laboratory samples, including Comprehensive Metabolic Panel (CMP), Complete Blood Count (CBC), Inflammatory Markers, and Coagulation panel.
* Physical examination by Principal Investigator.
* CHOP INTEND, PDMS-2 & PEDI-CAT by delegated personnel.

ELIGIBILITY:
Inclusion Criteria:

1. Subject diagnosed with LCMNA congenital muscular dystrophy.
2. Subject must have banked his stem cells at Hope Biosciences LLC.

Exclusion Criteria:

1. Subject has any active infection requiring medications.
2. The subject has any known coagulation anomalies.

Sex: All
Age Groups: Child, Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Djamchid Lotfi, MD, Principal Investigator — Investigator
Locations (1):
- Hope Biosciences Stem Cell Research Foundation, Sugar Land, Texas, United States